CLINICAL TRIAL: NCT06611241
Title: Hazard Anticipation Program for Parents of Teen Drivers
Acronym: HazAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth O'Neal (Other)
Responsible Party: Sponsor-Investigator, Elizabeth O'Neal, Assistant Professor, Community and Behavioral Health, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202010535
Record Dates: First submitted 2024-09-02; First posted 2024-09-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-02

CONDITIONS: Motor Vehicle Accident; Interaction, Parent-Offspring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hazard Anticipation Program for Parents of Teen Drivers (Experimental): Parents and teens randomly assigned to this arm of the trial will engage in a web-based training that provides parents with guidance on how to train their teen to identify potential hazards on the roadway. Parents are also given an opportunity to practice these new skills with teens when watching videos unfold together. The program will take 4 hours to complete and can be done over a two-week period at the parent's convenience.
  Interventions: Behavioral: Hazard Anticipation Program for Parents of Teen Drivers
- Control (No Intervention): The parents and teens in this arm of the study will not receive an intervention of any kind.

INTERVENTIONS:
Behavioral: Hazard Anticipation Program for Parents of Teen Drivers — Parents and teens who receive the intervention will complete a web-based training that provides parents with guidance on how to teach their teen to identify potential hazards on the roadway. The program begins by providing background on teens' difficulty learning this skill and the motivational interviewing techniques that are being used in the course. Parents then engage with a series of hazard videos. For each hazard, parents watch the hazard unfold, provide an example of what they might say to their teen in that, and are provided with examples of how to coach their teen through the hazard before it becomes a critical event. Parents and teens then jointly watch 12 videos depicting hazards unfolding on the roadway. Teens are asked to identify the hazard without parental input by pressing a spacebar. Teens must also indicate what they believe was the key event that caused the hazard. Then parents and teens are given an opportunity to replay the video and discuss the hazard together.
  Other Names: HazAPP
  Arms: Hazard Anticipation Program for Parents of Teen Drivers

SUMMARY:
This study will test an intervention that was developed to improve parents' driving instruction of teens' hazard anticipation skills when teens are in the learner phase of licensure. Half of the parents in the study will receive the intervention and half will not. Investigators will then compare driving instructions given by parents in the two groups by recording driving sessions that parents and teens have together in that real world and by recording a drive that parents and teens will complete in a driving simulator. The driving simulator allows us to expose teens and parents to hazards they may encounter on the roadway without putting them in harm's way.

DETAILED DESCRIPTION:
The project seeks to test an intervention designed to improve parents' communication about roadway hazards by comparing parent instruction and teen driving outcomes between dyads whose parents were assigned to the intervention vs. the control condition. Participants will be 100 parent-teen dyads. Half of the parent-teen dyads will receive the intervention and half will not. Parents who receive the intervention will complete web-based program developed to help parents instruct teens on how to identify hazards on the roadway and respond appropriately before they pose a crash risk. Parents in the intervention arm of the study will be given 2 weeks to complete the training. Parents in the control arm of the study will not receive training. After the delivery period, parents and teens will be given two additional weeks to apply the training in their everyday driving instruction. During this period, parents in both groups will complete a minimum of 5 drives with their teen that will be recorded. Investigators will then have teens and parents complete a drive in a driving simulator. Teens will drive and parents will instruct from the passenger seat, just like they would in the real world. The drive will have 12 hazards. Compared to parents in the control group, investigators believe that parents in the intervention group will exhibit improved communication about potential hazard detection with their teens. Similarly, the investigators believe that teens of parents who received the training will be better at anticipating and reacting to potential hazards on the roadway when driving independently compared to teens whose parents did not engage in the program.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents must be between the ages of 14 and 17 years. Additionally, they must be in the learner period of licensure.
* Parents must be the primary instructor of their teen's supervised driving.

Exclusion Criteria:

-

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-01-12 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Parental instruction of teen's driving in vehicle | Measures of parental instruction of teen's driving in the simulator will take place approximately between weeks 2 and 4 weeks of study enrollment.
  Investigators will code whether the parent verbally identifies the hazard, whether instruction from parents is functional or higher order in nature, and if instruction precedes or follows the hazard event. Functional instruction refers to instruction that applies only to the current context (e.g., "Slow down."). High-order instruction can be applied more generally to driving (e.g., "When there are brake lights ahead, be ready to brake too.") or why the hazard is dangerous by causally connecting dangerous features and their potential outcomes
Parental instruction of teen's driving in simulator | Measures of parental instruction of teen's driving in the simulator will take place approximately 4 weeks after enrollment.
  For the simulator drive, investigators will code whether the parent verbally identifies the hazard, whether instruction from parents is functional or higher order in nature, and if instruction precedes or follows the hazard event. Functional instruction refers to instruction that applies only to the current context (e.g., "Slow down."). High-order instruction can be applied more generally to driving (e.g., "When there are brake lights ahead, be ready to brake too.") or why the hazard is dangerous by causally connecting dangerous features and their potential outcomes
Teens driving performance in simulator - lane position | Measures of teen&#39;s driving performance in the simulator will take place approximately 4 weeks after enrollment.
  For the simulator driver investigators will also measure if parental instruction result in improved driving performance among teens. The investigators will specifically measure differences in lane position among the two groups in response to roadway hazards and parental instruction.

SECONDARY OUTCOMES:
Teens driving performance - accelerator release | Measures of teen&#39;s accelerator release in the simulator will take place approximately 4 weeks after enrollment.
  For the simulator driver investigators will also measure if parental instruction result in improved driving performance among teens. Investigators will specifically measure differences in accelerator release among the two groups in response to roadway hazards and parental instruction.
Teens driving performance in simulator - brake force | Measures of teen&amp;amp;#39;s driving performance in the simulator will take place approximately 4 weeks after enrollment.
  For the simulator driver investigators will also measure if parental instruction result in improved driving performance among teens. Investigators will specifically measure differences in lane position among the two groups in response to roadway hazards and parental instruction.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data that will program performance metrics (reaction time, accuracy). Data gathered during testing includes reduced metrics of simulator driving performance (speed, lane position, brake force, and acceleration), video capture of parent-teen interactions in naturalistic and simulated roadway environments, parent-teen interaction data reduced via reliable conversation coding, and questionnaire data reported by both parents and teens (e.g., family communication pattern, parenting style, teen temperament, assessment of the driving environment during driving sessions).
  Shared data will be de-identified and original data will be maintained at the primary investigator's institution. Video data will be deidentified to the extent possible.
  The investigators will archive all data, metadata, study protocols, and demonstration videos on Databrary (https://nyu.databrary.org/). Databrary is an NSF- and NIH-supported data sharing and archiving site, specializing in studies with children.
Supporting Information: Study Protocol, ICF
Time Frame: This information will be made available at the time of publication and will be available on Databrary in perpetuity.
Access Criteria: Anyone who receives IRB (or equivalent) approval can gain access tot the shared data.